CLINICAL TRIAL: NCT06357728
Title: Integrated Continuous Glucose Monitoring Glycemic cHAracterization During Pregnancy in Comparison With OGTT (I-CHAP)
Brief Title: Continuous Glucose Monitoring Glycemic cHAracterization During Pregnancy
Acronym: I-CHAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024/2035
Record Dates: First submitted 2024-03-18; First posted 2024-04-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-03

CONDITIONS: Gestational Diabetes; Glucose Metabolism Disorders; Metabolic Disease
Keywords: gestational diabetes; pregnancy; continuous glucose monitoring
MeSH Terms: conditions — Diabetes, Gestational; Glucose Metabolism Disorders; Metabolic Diseases | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: All participants will be given a continuous glucose monitoring device to wear for 10 days before during and after the oral glucose tolerance test.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous glucose monitoring arm (Experimental): Continuous glucose monitoring sensor: All study participants wear the sensor on the back of either right or left upper arm for up to 10 days. Glucose levels will be recorded from the interstitial fluid every 5 minutes using intermittent/ flash glucose scanning. Data will be captured using a receiver.
  Interventions: Device: Continuous glucose monitoring

INTERVENTIONS:
Device: Continuous glucose monitoring — Continuous glucose monitoring sensor: All study participants wear the sensor on the back of either right or left upper arm for up to 10 days. Glucose levels will be recorded from the interstitial fluid every 5 minutes using intermittent/ flash glucose scanning. Data will be captured using a receiver.

SUMMARY:
Our study named Integrated Continuous glucose monitoring glycemic cHAracterization during Pregnancy in comparison with oral glucose tolerance test (I-CHAP) aims to establish much needed preliminary evidence in our Asian population to show the capabilities of CGM use and its wealth of data for GDM diagnosis. This study aims to test the following aims and hypotheses in a single-armed intervention pilot trial study of pregnant women undergoing the oral glucose tolerance test:

Aim 1. To characterize CGM glucose values with the 3-point blood glucose measured during the OGTT procedure.

The investigators hypothesize that the CGM glucose values at single time points while fasted, and after the 75-g glucose load will be positively correlated with 3-timepoint blood glucose values captured during the OGTT.

Aim 2. To correlate the CGM glucose excursions and CGM-derived metrics (glycaemic variability and glycaemic control) with maternal-fetal outcomes and treatment outcomes.

The investigators hypothesize that higher AUC, glycemic variability and poorer glycaemic control will better distinguish maternal-fetal outcomes and treatment outcomes, compared to the OGTT.

Aim 3. To describe the acceptability of using the Dexcom G6 CGM as a diagnostic tool instead of the OGTT. The investigators hypothesize that a higher proportion of participants will report CGM to be more acceptable than the OGTT for GDM diagnosis.

DETAILED DESCRIPTION:
This proposal aims to address one of Singapore's major clinical challenges, which is the very high prevalence of GDM, and the current approach to GDM diagnosis. With the current practices, guidelines by the IADPSG, as well as the Singaporean guidelines recommend universal screening of GDM among all pregnant women at 24-28 weeks of gestation, which reveals the very high prevalence of GDM with 20-25% diagnosed by mid-pregnancy. The precision in GDM monitoring and treatment is important not only for the short-term adverse outcomes related to pregnancy and delivery, but as local studies have shown, also for the long-term consequences affecting both the mother and the child such as development of Type II Diabetes (T2D), obesity, metabolic, cardiovascular, neurodevelopment and psychiatric problems. While many patients can reach their target glucose levels through lifestyle behavior adjustments (diet and exercise), around 30% may require pharmacological interventions. Additionally, even individuals with only slightly elevated glucose levels, who don't meet the typical GDM criteria could experience better pregnancy outcomes if treated. This is because the connection between glucose levels and adverse pregnancy outcomes, such as macrosomia, remains consistent across a range of increasing glucose levels.

The primary gap in current research lies in the exploration of CGM use during pregnancy for diagnosing GDM, with the aim of leveraging the distinctive CGM glucose profiles to predict adverse maternal-fetal outcomes and advocate for a revised treatment approach. As CGM usage becomes increasingly accepted in clinical practice, there is a growing need for further research to advance this technology and explore the optimal ways to utilize the data it produces for improved GDM diagnosis and treatment strategies.

In this pilot single-arm intervention study, 60 pregnant women of only Chinese or Indian ethnicity with a GDM rate of 20% will be recruited from the KK Women's and Children's Hospital (KKH) outpatient obstetrics and gynaecology clinic. The participants recruited before scheduled OGTT's will be educated on how to put on the CGM after completing a consent form. Participants will be educated on how to put on the CGM device before their scheduled OGTTs at 20-35 weeks as an acclimation period and will undergo the OGTT before CGM removal on the 10th day of wear. Patients will be told to record the exact date and time of the OGTT. Exclusion criteria were pre-existing Type 1 or Type 2 diabetes, mental illness precluding informed consent and women who were diagnosed early (1st or early 2nd trimester for GDM).

Data will be collected through questionnaires and a case report form. The questionnaires include socio-economic factors, and baseline characteristics. The case report form will be collecting data on the OGTT glucose test results, as well as maternal obstetrics and birth outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women of only Chinese or Indian ethnicity
2. Pregnant women between age 21--45 years old
3. Oral glucose tolerance test (OGTT) to be scheduled between 20-35 weeks gestational age
4. OGTT to be done at KK Women's and Children's Hospital

Exclusion Criteria:

1. Women with serious skin conditions (e.g. eczema) that precludes wearing the sensor for 10 days
2. Exclusion criteria were pre-existing Type 1 or Type 2 diabetes, mental illness precluding informed consent and women who were diagnosed early (1st or early 2nd trimester for GDM).

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Maternal plasma glucose values measured by oral glucose tolerance test (OGTT) at 0-hour (mmol/L) | During OGTT procedure at 20-35 weeks gestation
  Three-point OGTT (fasting, 1-hour and 2-hour) will be performed at 20-35 weeks gestation
Maternal plasma glucose values measured by oral glucose tolerance test (OGTT) at 1-hour (mmol/L) | During OGTT procedure at 20-35 weeks gestation
  Three-point OGTT (fasting, 1-hour and 2-hour) will be performed at 20-35 weeks gestation
Maternal plasma glucose values measured by oral glucose tolerance test (OGTT) at 2-hour (mmol/L) | During OGTT procedure at 20-35 weeks gestation
  Three-point OGTT (fasting, 1-hour and 2-hour) will be performed at 20-35 weeks gestation

SECONDARY OUTCOMES:
Maternal obstetric outcomes - Pre-eclampsia | At the end of pregnancy at 40-42 weeks
  Pre-eclampsia will be retrieved from medical notes after delivery
Maternal obstetric outcomes- Pregnancy-induced hypertension | At the end of pregnancy at 40-42 weeks
  Pregnancy-induced hypertension will be retrieved from the medical notes after delivery
Maternal obstetric outcomes - C-section | At the end of pregnancy at 40-42 weeks
  C-section delivery will be retrieved from the medical notes after delivery
Neonatal outcomes- Large-for-gestational-age | At the end of pregnancy at 40-42 weeks
  Large-for-gestational-age will be retrieved from the medical notes after delivery.
Neonatal outcomes-Birth weigh | At the end of pregnancy at 40-42 weeks
  Birth weight will be retrieved from the medical notes after delivery.
Neonatal outcomes- Small-for-gestational-age | At the end of pregnancy at 40-42 weeks
  Small-for-gestational-age will be retrieved from the medical notes after delivery.
Neonatal outcomes-Pre-term birth | At the end of pregnancy at 40-42 weeks
  Pre-term birth will be retrieved from the medical notes after delivery.
Neonatal outcomes-Neonatal hypoglycaemia | At the end of pregnancy at 40-42 weeks
  Neonatal hypoglycaemia will be retrieved from the medical notes after delivery.

OTHER OUTCOMES:
Types of treatment received for gestational diabetes diagnosis | At the end of pregnancy at 40-42 weeks
  Type of treatment (i.e diet only, insulin, or diet and metformin) received by study participants will be recorded from medical notes after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Phaik Ling, Elaine Quah, PhD, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT06357728/Prot_SAP_ICF_000.pdf